CLINICAL TRIAL: NCT05193929
Title: A Multi-center, Randomized Controlled Clinical Investigation Evaluating Wound Closure with OptiPulse™ Versus Standard of Care in the Treatment of Non-Healing Diabetic Foot Ulcers
Brief Title: A Clinical Investigation Evaluating Wound Closure with OptiPulse™ Versus SOC in the Treatment of Non-Healing DFU's
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Compedica Inc (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBC-PUL-02
Record Dates: First submitted 2021-12-13; First posted 2022-01-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OptiPulse™ (Experimental): The OptiPulse™ is designed to enhance blood circulation in the venules and arterioles in subjects with diabetic foot ulcers of the lower extremities. OptiPulse™ is supplied as a pair of footwear. One side is fitted with an offloaded and shin pumping unit and the other acts as pressure reducing footwear. Both active and non-active footwear should be worn to give balanced gait.
  Interventions: Device: OptiPulse™
- Standard of care offloading device (Active Comparator): Diabetic CAM boot
  Interventions: Device: Standard of Care offloading device

INTERVENTIONS:
Device: OptiPulse™ — TheOptiPulse™ is designed to enhance blood circulation in the venules and arterioles in subjects with diabetic foot ulcers of the lower extremities. OptiPulse™ is supplied as a pair of footwear. One side is fitted with an off loader and shin pumping unit, and the other acts as pressure reducing footwear.Both active and non-active footwear should be worn to give balanced gait
  Arms: OptiPulse™
Device: Standard of Care offloading device — CAM boot
  Arms: Standard of care offloading device

SUMMARY:
The purpose of this clinical investigation is to assess the safety and performance of Compedica's OptiPulse™ and to collect subject outcome data on the treatment of diabetic foot ulcers (DFU's) versus the standard of care (SOC). OptiPulse™ is designed to enhance blood circulation in the venules and arterioles. Fibracol Plus (or equivalent) is a collagen alginate dressing that is used as the primary dressing. Both products are 510(k) FDA cleared and will be used within the cleared intended use.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old, inclusive.
2. Presence of a DFU, Wagner Grade 1 (see Appendix A for definitions) on the plantar or dorsal aspect of the foot, extending through the dermis provided it is below the medial aspect of the malleolus.
3. The index ulcer will be the largest ulcer if two or more DFUs are present with the same Wagner grade and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
4. Index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to SV1 and less than 1 year, as of the date the subject consents for study.
5. Index ulcer is a minimum of 0.8 cm2 and a maximum of 25 cm2 at SV1 and TV1.
6. Within 3 months of SV1, adequate circulation to the affected foot, as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) between 0.7 and 1.3 within 3 months of SV1, using the affected study extremity. As an alternative arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of > 0.6 is acceptable.
7. The target ulcer has been offloaded for at least 14 days prior to randomization.
8. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
9. Subject understands and is willing to participate in the clinical study and can comply with weekly visits.
10. Subjects must have read and signed the IRB approved ICF before screening procedures are performed.

Exclusion Criteria:

* 1. Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.

  2. Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.

  3. Index ulcer is overtly infected (i.e. purulent drainage). 4. Subjects with a history of more than two weeks of treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study.

  5. Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1.

  6. History of radiation at the ulcer site (regardless of time since last radiation treatment).

  7. Index ulcer has been previously treated or will need to be treated with any prohibited therapies.

  8. Subjects with a previous diagnosis of HIV or Hepatitis C. 9. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.

  10. Osteomyelitis or bone infection of the affected foot as verified by x-ray within 30 days prior to the first screening visit. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).

  11. Subject is pregnant or breast-feeding. 12. Presence of diabetes with poor metabolic control as documented with an HbA1c >12.0 within last 90 days.

  13. Subjects with end-stage renal disease as evidenced by a serum creatinine ≥3.0 mg/dL within 6 months of randomization. 14. Presence of active Charcot Neuroarthropathy to the affected limb. 15. Any wound located entirely on the medial or lateral border of the foot. 16. Any wound located between the 1st through 4th toe interspaces. 17. Index ulcer has reduced in area by 30% or more after 14 days of SOC from SV1 to the TV1/Randomization visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of index ulcers healed | 12 weeks

SECONDARY OUTCOMES:
Time to Ulcer Healing | 12 weeks
Percentage Area Change | 6 and 12 weeks
Changes in wound quality of life from screening visit to end of study ( per W-QoL) | 12 weeks

OTHER OUTCOMES:
Cost to Closure | 12 weeks

CONTACTS AND LOCATIONS:
Locations (19):
- United States (18):
  - Titan Clinical Research, Phoenix, Arizona
  - Felix Sigal, Los Angeles, California
  - Clemente Clinical Research, Los Angeles, California
  - ILD Research, Vista, California
  - Midland Florida clinical Research Center LLC, DeLand, Florida
  - Integral Clinical Trial Solutions, Homestead, Florida
  - Integral Clinical Trials Solutions, Pembroke Pines, Florida
  - Integral Clinical Trials Solutions, Tamarac, Florida
  - Viable Research Management, Las Vegas, Nevada
  - Foot Associates of New York, New York, New York
  - Foot & Ankle specialists of the Mid-Atlantic, Gastonia, North Carolina
  - Foot & Ankle Specialists of the Mid-Atlantic, Raleigh, North Carolina
  - Lower Extremity Institution of Research and Therapy (LEIRT), Boardman, Ohio
  - Mt. Olympus Medical Research, Houston, Texas
  - Clinical Trials Network, Houston, Texas
  - Foot and Ankle Specialist of the Mid-Atlantic - Roanoke, Roanoke, Virginia
  - Foot and Ankle Specialist of the Mid-Atlantic - Salem, Salem, Virginia
  - Salem Research institute, Salem, Virginia
- East Toronto Vascular Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No